CLINICAL TRIAL: NCT04021225
Title: A Multicenter, Randomized, Controlled Study According to §23b Medical Devices Act (MPG) Comparison of Ectoin® Eyedrops & Ectoin® Eye Spray With Tears Again® for the Application of Environmental Disorders of the Eye of Allergic Patients.
Brief Title: Comparison of Ectoin® Containing Eye Drops and Ectoin® Containing Eye Spray With the Eye Spray Tears Again®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: btph-015-2018-AAT04-EES09
Record Dates: First submitted 2019-05-07; First posted 2019-07-16 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Eye Manifestations
Keywords: According to section 23b Medical Devices Act; environmental disorder eye; allergen exposure; Ectoin® Allergy Eye Drops 2%; Ectoin® Eye Spray Colloidal; Ectoin
MeSH Terms: conditions — Eye Manifestations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ectoin® Allergy Eye Drops 2% (Active Comparator): 20 Patients:
  - Ectoin® Allergy Eye Drops 2% (bitop AG)
  Interventions: Device: Ectoin® Allergy Eye Drops 2%
- Ectoin® Eye Spray Colloidal (Active Comparator): 20 Patients:
  -Ectoin® Eye Spray Colloidal (bitop AG)
  Interventions: Device: Ectoin® Eye Spray Colloidal
- Tears Again® Eye Spray (Active Comparator): 20 Patients:
  - Tears Again® Eye Spray (Optima Pharmazeutische GmbH)
  Interventions: Device: Tears Again® eye spray

INTERVENTIONS:
Device: Ectoin® Allergy Eye Drops 2% — A one-time application of 1-2 drops in the more affected eye will be investigated.
  Arms: Ectoin® Allergy Eye Drops 2%
Device: Ectoin® Eye Spray Colloidal — A one-time application of 1-2 drops in the more affected eye will be investigated.
  Arms: Ectoin® Eye Spray Colloidal
Device: Tears Again® eye spray — A one-time application of 1-2 drops in the more affected eye will be investigated.
  Arms: Tears Again® Eye Spray

SUMMARY:
This study aims to gain knowledge on the duration of symptom relief of environmental disorders of the eye as might be present in allergy sufferers after allergen exposure following application of the study products.

Additionally, the extent of symptom relief as well as tolerability of this topic treatment will be evaluated.

DETAILED DESCRIPTION:
The term disorder describes the general development of physical symptoms without vegetative or morphologically detectable impairment.

These disorders cause physical symptoms with different severities and different impairments, e.g. exhaustion, fatigue, headache, stomach and back pain.

The eye might also be prone to disorders. These manifest in symptoms like dry eyes, tightness of the eye lids, foreign body sensation and reddened, burning, itching or watery eyes.

Disorders of the eye can be caused by extensive screen and computer work, air condition, dry heating air or draught, as well as some drugs like birth control pills, or beta blocker. Other causes are intense solar radiation or allergen exposure.

To reduce the symptoms, medical products like artificial tears (with fat additives, if necessary, and applied as drops, gel or spray) are used to moisten the eyes and the eye lids. Besides, eye drops and eye sprays (with different supplements) are also used to stabilise the tear film.

The positive effect of Ectoin® was already proven in many studies: Ectoin® containing products exhibited a good barrier function and effective protection against dehydration of the skin.

Another formulation of Ectoin® for the use on the eye is Ectoin® Eye Spray Colloidal. This spray is - in analogy to Tears Again® eye spay - applied to the closed eye lids and moistens the surface of the eye with an Ectoin® containing liquid film after opening the eye.

This form of application of Ectoin® is also registered as a medical product for dry, irritated and inflamed eyes as well as the adjacent skin.

Ectoin® Allergy Eye Drops 2% protect against harmful influences of allergens and support the regeneration of irritated and sensitive conjunctiva.

The package leaflet recommends the application of 1-2 drops in each eye several times a day. In the scope of this study, a one-time application of 1-2 drops in the more affected eye will be investigated.

Ectoin® Eye Spray - Colloidal moistens the eye and thus protects the eye against hyperosmolarity of the tear fluid. The package leaflet recommends the application of 1-2 sprays on the closed eye 3-4 times a day. In the scope of this study, a one-time application of 1-2 sprays in the more affected eye will be investigated.

Tears Again® is a liposomal eye spray, which stabilises the lipid layer of the tear film and thus improves the moistness of the surface of the eye: the underlying tear fluid is protected against quick evaporation or against flow off the lid edge. The summary of product characteristics recommends the application of 1-2 sprays on the closed eye up to 3-4 times a day. A more frequent application, especially in cases of severe disorders is possible without any problems. Within the current study, a on-time application of 1-2 sprays to the more affected eye will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Patients have to meet the following inclusion criteria in order to participate in the study:

* Signed and dated informed consent form
* Male and female patients aged 18 to 75 years
* Patients have to suffer from allergen exposure induced environmental disorder of the eye

Exclusion Criteria:

-

Non-inclusion criteria

* Contraindications according to the package leaflet/summary of product characteristics
* currently wearing contact lenses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Patient questionnaire | Change is being assessed between before the application of the medical product and 30 minutes after the application of the medical product.
  Relief of environmental disorders of the eye will be assessed by determining the time to onset of action using a patient questionnaire. The extent of relief as the degree of effectiveness will be determined using the following variables:
  • Patient questionnaire
  The questions from the patient questionnaire are:
  * How do you rate your eyesight at this time? Unimpaired, impaired
  * Do you have difficulties reading normal printed material in the newspaper? (no, a little, strong, stopped trying)
Assessment of the redness of the eye | Change is being assessed between before the application of the medical product and 30 minutes after the application of the medical product.
  Relief of environmental disorders of the eye will be assessed by determining the time to onset of action using a patient questionnaire. The extent of relief as the degree of effectiveness will be determined using the following variables:
  • Digital analysis of the redness of the eye.
  The redness of the eye is evaluated by means of digital image analysis. The patient's more affected eye is photographed parallel to the entries on the VAS. To capture the images, the same construction for attaching the camera as well as fixed camera settings are used to create comparable conditions. Captured data analyzed by MATLAB V.9.5.
Assessment of the redness of the eye by an external observer | Change is being assessed between before the application of the medical product and 30 minutes after the application of the medical product.
  Relief of environmental disorders of the eye will be assessed by determining the time to onset of action using a patient questionnaire. The extent of relief as the degree of effectiveness will be determined using the following variables:
  • Assessment of the redness of the eye by an external observer
  Redness of eye evaluated by a physician.
Visual Analogue Scale | Change is being assessed between before the application of the medical product and 30 minutes after the application of the medical product.
  Relief of environmental disorders of the eye will be assessed by determining the time to onset of action using a patient questionnaire. The extent of relief as the degree of effectiveness will be determined using the following variables:
  • Visual Analogue Scale
  The evaluation of effectiveness data is collected by the patient using a visual analogue scale. To this end, the patient marks on a visual analog scale by a vertical line the extent of his discomfort between the endpoints most severe complaints = 100 and no complaints = 0.
Tolerability: The degree of irritation of the tested eye is being measured using a visual analogue scale. | Change is being assessed between 0 minutes and 30 minutes after the application of the medical product.
  It will be assessed using the following variables:
  • The patient questionnaires are:
  Please evaluate the degree of irritation of the tested eye (itching, foreign body sensation, lacrimation and/or swelling of the eyelid) after administration of the investigational medicinal product.
  The evaluation of effectiveness data is collected by the patient using a visual analogue scale. To this end, the patient marks on a visual analog scale by a vertical line the extent of his discomfort between the endpoints most severe complaints = 100 and no complaints = 0.
Safety: All adverse reactions and adverse events that occur after signing the informed consent form must be reported, even if no investigational medicinal product was taken. | Up to 12 hours after the application of medical product.
  It will be assessed using the following variables:
  • The occurrence of adverse events.
  Safety: Adverse events and serious adverse events evaluated by physicians. Any side effects that were not present before the visit, and any side effects that reoccur or worsen after the visit. Abnormal clinically relevant results from diagnostic procedures, including out-of-range laboratory testing, should be considered as an AE. If adverse reactions occur after the visit, the patient is encouraged to contact the doctor by telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, Dr., Study Director — ClinCompetence
Locations (1):
- Facharzt für HNO-Heilkunde, Allergologie, Aachen, North Rhine-Westphalia, Germany